CLINICAL TRIAL: NCT01769248
Title: Randomized Prospective Trial of EUS-FNA Versus EUS-FNB Using a Novel Core Biopsy Needle
Brief Title: Prospective Trial of EUS-FNA Versus EUS-FNB Using a Novel Core Biopsy Needle
Acronym: MUCIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Sri Komanduri, Associate Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: FNAFNBmucin
Record Dates: First submitted 2013-01-10; First posted 2013-01-16 (Estimated); Results first posted 2015-03-18 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2017-12

CONDITIONS: Pancreatic Cancer; Lymphadenopathy; Gastrointestinal Stromal Tumor
Keywords: EUS; FNA; FNB
MeSH Terms: conditions — Pancreatic Neoplasms; Lymphadenopathy; Gastrointestinal Stromal Tumors | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fine needle aspiration (Active Comparator): fine needle aspiration
  Interventions: Device: Fine needle aspiration; Device: Fine needle biopsy
- Fine needle biopsy (Active Comparator): Fine needle biopsy
  Interventions: Device: Fine needle aspiration; Device: Fine needle biopsy

INTERVENTIONS:
Device: Fine needle aspiration — Fine needle aspiration
  Other Names: Echo Tip FNA Needle
Device: Fine needle biopsy — FNB
  Other Names: Echo Tip Procore

SUMMARY:
Endoscopic ultrasound (EUS) is paramount in the diagnosis and evaluation of cancers involving the gastrointestinal tract. EUS allows for the acquisition of cellular (fine needle aspirate - FNA) or tissue biopsy (fine needle biopsy - FNB) for diagnostic purposes. This has traditionally been done with fine needle aspirate where a needle is inserted into the tumor and potentially malignant cells are extracted for microscopic analysis. More recently, a needle that allows a tissue biopsy for histologic analysis has been FDA approved.

The Echotip Procore (Cook Medical) core biopsy needle (ETP), has been demonstrated to provide excellent efficacy for core biopsy samples. Final diagnostic yield using this needle ranges from 80-90% and appears to be significantly greater than EUS-FNA for lesions requiring histology for diagnosis. However, there is currently only limited data from prospective studies comparing EUS-FNA to EUS-FNB with the ETP needle. The investigators propose a randomized, prospective, cross-over study comparing diagnostic accuracy of EUS-FNA to EUS-FNB.

DETAILED DESCRIPTION:
Endoscopic ultrasound (EUS) is paramount in the diagnosis and evaluation of cancers involving the gastrointestinal tract. EUS allows for the acquisition of cellular (fine needle aspirate - FNA) or tissue biopsy (fine needle biopsy - FNB) for diagnostic purposes. This has traditionally been done with fine needle aspirate where a needle is inserted into the tumor and potentially malignant cells are extracted for microscopic analysis. More recently, a needle that allows a tissue biopsy for histologic analysis has been FDA approved.

We will compare tissue samples obtained by standard FNA to FNB with a sample size of 140 patients with the primary outcome being diagnostic yield. Each patient will be randomized to FNA or FNA. If after 3 passes the on-site evaluation remains inadequate, the endoscopist will crossover to the other arm.

ELIGIBILITY:
Inclusion Criteria:

- 3.1.1 All patients referred for EUS tissue sampling who provide informed consent

Exclusion Criteria:

* 3.2.1 Coagulopathy which is not corrected

3.2.2 Diagnostic EUS determines lesion is not amenable to FNA or FNB

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinadh Komanduri, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - UCLA Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Moffit Cancer Center, Tampa, Florida

RESULTS

PARTICIPANT FLOW:
Groups:
- Fine Needle Aspiration (FNA): fine needle aspiration
  Fine needle aspiration: Fine needle aspiration using endoscopic ultrasound-FNA needles. This was the standard of care arm
- Fine Needle Biopsy (FNB): Fine Needle biopsy
  Fine Needle biopsy: FNB, test arm for core biopsies, endoscopic ultrasound-FNB
Period: Overall Study
Arm/Group | Fine Needle Aspiration (FNA) | Fine Needle Biopsy (FNB)
Started | 70 | 70
Participants Who Crossed-over | 28 | 12
Completed | 42 | 58
Not Completed | 28 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fine Needle Aspiration | Fine Needle Biopsy | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 57 | 107
  >=65 years | 20 | 13 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (14.4) | 64.1 (14.4) | 63.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 30 | 66
  Male | 34 | 40 | 74
Region of Enrollment [Number; unit: participants]
  United States | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Yield of EUS-FNB and EUS-FNA
Description: The investigators' primary outcome measure will assess the diagnostic yield (percentage of patients with a diagnosis) of EUS-FNB (fine-needle biopsy) to provide a final diagnosis of the lesion being sampled. This will be expressed as a percentage.
Time Frame: 1 year
Measure: Number; unit: percentage of patients
Arm/Group | Fine Needle Aspiration | Fine Needle Biopsy
Number analyzed (Participants) | 70 | 70
percentage of patients | 67.1 | 90

2. Secondary Outcome: Specimen Adequacy as Assessed by Rapid-onsite Evaluation of FNA and FNB
Description: The investigators' secondary outcome will assess the ability to obtain an adequate specimen for in room cytologic evaluation as determined by our cytopathologist. This will be defined as a sample that is representative (not necessarily diagnostic) of the lesion in question. This will be expressed as a percentage and compared between FNA and FNB
Time Frame: 1 year
Population: Patients with pancreatic and non-pancreatic lesions receiving EUS-FNA and EUS-FNB.
Measure: Number; unit: percentage of participants
Arm/Group | Fine Needle Aspiration | Fine Needle Biopsy
Number analyzed (Participants) | 70 | 70
percentage of participants | 60.0 | 82.8

3. Secondary Outcome: Percentage of Patients in Whom a Diagnosis is Achieved After Crossover (%)
Description: As above. Crossover to FNA or FNB occurs after 3 passes without adequate material
Time Frame: 1 yr
Population: Participants receiving alternative tissue acquisition method when initial three passes with either EUS-FNA or EUS-FNB failed to provide an adequate specimen.
Measure: Number; unit: percentage of participants
Groups:
- Fine Needle Aspiration to Fine Needle Biopsy: fine needle aspiration to fine needle biopsy
  EUS-FNA to EUS-FNB
- Fine Needle Biopsy to Fine Needle Aspiration: Fine needle biopsy to fine needle aspiration
  EUS-FNB to EUS-FNA
Arm/Group | Fine Needle Aspiration to Fine Needle Biopsy | Fine Needle Biopsy to Fine Needle Aspiration
Number analyzed (Participants) | 28 | 12
percentage of participants | 96.4 | 41.7

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Fine Needle Aspiration | Fine Needle Biopsy
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No